CLINICAL TRIAL: NCT02957461
Title: Validation of Brain Function Assessment Algorithm for mTBI From Injury to Rehabilitation in College Athletes
Brief Title: Validation of Brain Function Assessment Algorithm for mTBI/Concussion in College Athletes
Acronym: CASVAL
Status: Completed | Type: Observational
Sponsor: BrainScope Company, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 18-Ahead
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2018-08

CONDITIONS: Brain Injuries, Traumatic; Concussion, Mild; Concussion, Brain; Concussion, Severe; Concussion, Intermediate
Keywords: Concussion; Mild Traumatic Brain Injury; Sport Related Concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Injured and Matched Control Subject Pool: Injured subjects consist of athletes who are head injured and meet the inclusion/exclusion criteria. Injured subjects will be tested within 72 hours (3 days) of injury and at specified time points post injury. Matched control subjects will be tested at the same time intervals as the injured subject. BrainScope Battery will be performed at each time point and consists of the following components: brain electrical activity (EEG), neurocognitive performance assessment, ocular motor assessment, and clinical symptoms/assessments.
  Interventions: Device: BrainScope Ahead 200iD
- Healthy Volunteer Subject Pool: This subject pool will consist of uninjured (not head injured) contact and non-contact athletes and will be tested at a single time point. These subjects will perform the same BrainScope Battery as the injured and matched control subjects.
  Interventions: Device: BrainScope Ahead 200iD

INTERVENTIONS:
Device: BrainScope Ahead 200iD — The BrainScope Battery evaluation will consist of 4 tests to aid in the assessment of concussion: History, Physical, signs and symptoms (SAC, SCAT3), Electrophysiological Function; Neurocognitive Performance Assessment and Ocular Motor assessment. BrainScope Ahead 200iD device will be used to perform EEG.

SUMMARY:
This study is Part 1 of data collection from 18-25 years old subject population for validation of previously derived algorithms. This data will be combined with that collected under NCT03671083 (Part 2 with subject age range 13-25 years) for the final analyses of validation of the algorithms.

DETAILED DESCRIPTION:
EEG, neurocognitive performance and clinical data will be collected at time of injury (within 3 days) at clinically determined Return to Play (RTP) and 45 days after RTP, for the purpose of independently validating the performance of the algorithms developed in prior studies (NCT02477943, NCT02661633 and NCTXXXXXX). Data collected under this study will be combined with that collected under NCT03671083 for the final analyses of prospective algorithm performance in an independent population ages 13-25 years. Subjects will come from the sports and other populations of concussed individuals. They will be matched with controls i.e. not head injured subjects who will also undergo the same set of tests and the same time intervals as the injured subjects. An additional pool of uninjured (not head injured) subjects will be collected who will be assessed at a single time point.

ELIGIBILITY:
Inclusion Criteria (For Injured Subjects):

1. Time of injury within 72 hours of BrainScope Battery
2. No evidence of abnormality visible on Computerized Tomography (CT) of the head related to the traumatic event (Note: neuroimaging is not required for enrollment)
3. No hospital admission due to either head injury or collateral injuries for >24 hours
4. GCS between 13-15

Exclusion Criteria:

1. Previously enrolled as an Injured or Matched Control subject in the BrainScope Algorithm Development Study
2. Current CNS active prescription medications taken daily, with the exception of medications being taken for the treatment of Attention Deficit Disorder (ADD) or Attention Deficit Hyperactivity Disorder (ADHD)
3. Forehead, scalp or skull abnormalities that prevents headset application or EEG data collection
4. History of brain surgery or neurological disease
5. Pregnant women
6. Do not speak or read English
7. Loss of consciousness ≥ 20 minutes related to the concussion injury - for injured subjects only
8. Prior history of concussion in the last year - for Matched Control subjects only

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Approximately 220 male and female student-athletes from participating universities or colleges will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Likelihood of being concussed | 6 months for data acquisition, with each patient studied from time of injury to 45 days after RTP
  Sensitivity and specificity forthe identification of the likelihood of concussion/mTBI at the time of injury using a multi-modal EEG-based Concussion Index (CI)

SECONDARY OUTCOMES:
Significance of change over time | 6 months for data acquisition, with each patient studied from time of injury to 45 days after RTP
  Significant difference in concussion index between time of injury and return to play (RTP)
Prediction of prolonged recovery | 6 months for data acquisition, with each patient studied from time of injury to 45 days after RTP
  Accuracy of prediction of prolonged recovery from injury assessment using a multi-modal EEG-based concussion index

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Prichep, Ph.D., Study Director — BrainScope Company, Inc.
Locations (8):
- United States (8):
  - University of Arkansas, Fayetteville, Arkansas
  - University of Connecticut, Storrs, Connecticut
  - University of South Florida, Tampa, Florida
  - Michigan State University, East Lansing, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of South Carolina, Columbia, South Carolina
  - University of Texas - Austin, Austin, Texas